CLINICAL TRIAL: NCT05194514
Title: Randomized Trial to Compare the SherpaPak™ Device vs Cold Storage of Donor Hearts in Transplantation: A Pilot Study
Brief Title: Trial to Compare the SherpaPak™ Device vs Cold Storage
Acronym: SherpaPak
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Fardad Esmailian, Professor of Surgery, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00001753
Record Dates: First submitted 2021-12-23; First posted 2022-01-18 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Organ Transplant
MeSH Terms: interventions — Cryopreservation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SherpaPak™ Cardiac Transport System (Other): When a matching donor heart from a non-local donor offer (from Northern California, Arizona, Nevada or farther geographies) becomes available the recipient will be assigned a subject identification number and randomized 1:1 to receive a heart transported using either standard of care cold storage or the SherpaPak™ Cardiac Transport System.
  Interventions: Device: SherpaPak™ Device
- Cold Storage (Other): When a matching donor heart from a non-local donor offer (from Northern California, Arizona, Nevada or farther geographies) becomes available the recipient will be assigned a subject identification number and randomized 1:1 to receive a heart transported using either standard of care cold storage or the SherpaPak™ Cardiac Transport System.
  Interventions: Other: Cold Storage

INTERVENTIONS:
Device: SherpaPak™ Device — The SherpaPak™ Cardiac Transport System has been developed to provide a safe, consistent method for cold ischemic storage of donor hearts for transplantation. This device is FDA approved.
  Arms: SherpaPak™ Cardiac Transport System
Other: Cold Storage — FDA-approved method for organ procurement
  Arms: Cold Storage

SUMMARY:
The Investigator's are doing this study to see which method of organ preservation leads to better outcomes for donated hearts.

There are two methods of organ preservation. The first method is the use of cold storage. With this method, the donor heart is stored in preservation fluid within bags that are then placed on ice and transported in a cooler. This is the usual method for transporting donor hearts. This is also known as "standard of care."

The second method is the use of the SherpaPak™ Cardiac Transport System. With this method, the donor heart is kept at a steady, consistent temperature throughout transportation. This method is not typically used for transporting donor hearts.

The study will include up to 20 people in total.

DETAILED DESCRIPTION:
This is a randomized study and has 2 study groups. Participants will be randomly assigned to a group in a 1:1 ratio.

* 50% chance of receiving a donor heart using the SherpaPak™ method, or
* 50% chance of receiving a donor heart using the cold storage method.

The research team will analyze data from the medical records from the heart transplant and clinic visits up to 30 days after the heart transplant. Participants will be in the study for about 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Any sex/gender, 18 years of age or older listed for primary heart transplant.
* Subjects must be willing and be capable of understanding the purpose and risks of the study and must sign a statement of informed consent OR consent of a legally authorized representative of a cognitively impaired individual will be obtained before the cognitively impaired individual may be included in research.
* Signed: 1) written informed consent document and 2) authorization to use and disclose protected health information
* Subjects must receive and accept a non-local donor offer (from Northern California, Arizona, Nevada or farther geographies)

Exclusion Criteria:

* Re-do heart transplant
* Multi-organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fardad Esmailian, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data that underlies the results reported in this article, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: 1 year after the study is closed.
Access Criteria: Researchers who provide a methodologically sound proposal.

RESULTS

PARTICIPANT FLOW:
Groups:
- Cold Storage: Subjects that received donor hearts preserved with cold storage
- SherpaPak: Subjects who received donor hearts preserved through SherpaPak
Period: Overall Study
Arm/Group | Cold Storage | SherpaPak
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline Demographics for Recipient Standard Care Cold Storage: Standard Care Cold Storage
- Baseline Demographics for Recipient Sherpapak: Baseline demographics for recipient Standard Care Cold Storage
- Total: Total of all reporting groups
Arm/Group | Baseline Demographics for Recipient Standard Care Cold Storage | Baseline Demographics for Recipient Sherpapak | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 62 (9.3) | 57.2 (9.7) | 59.7 (9.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex (male) | 6 | 8 | 14
  Sex (female) | 4 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity (non-hispanic) | 6 | 5 | 11
  Ethnicity (hispanic) | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Absence of Moderate to Severe Primary Graft Dysfunction (Left or Right Ventricle)
Description: Percentage of subjects without moderate to severe primary graft dysfunction (left or right ventricle)
Time Frame: 24 hours post-transplant
Measure: Count of Participants; unit: Participants
Groups:
- Standard Care Cold Storage; Sherpapak Cardiac Transport: 100% freedom from severe primary graft dysfunction
Arm/Group | Standard Care Cold Storage | Sherpapak Cardiac Transport
Number analyzed (Participants) | 10 | 10
Participants | 10 | 10

2. Primary Outcome: 30-day Post-transplant Survival
Time Frame: 30 day post heart transplant (htx)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care Cold Storage | Sherpapak Cardiac Transport
Number analyzed (Participants) | 10 | 10
Participants | 10 | 9

3. Primary Outcome: Freedom From 30-day Ischemic Reperfusion Injury
Time Frame: 30 day post htx
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care Cold Storage | Sherpapak Cardiac Transport
Number analyzed (Participants) | 10 | 10
Participants | 10 | 8

4. Primary Outcome: Freedom From 30-day Biopsy Proven Rejection
Time Frame: 30 day post htx
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care Cold Storage | Sherpapak Cardiac Transport
Number analyzed (Participants) | 10 | 10
Participants | 9 | 8

5. Primary Outcome: Freedom From 30-day Any-treated Rejection
Time Frame: 30 day post htx
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care Cold Storage | Sherpapak Cardiac Transport
Number analyzed (Participants) | 10 | 10
Participants | 9 | 8

6. Secondary Outcome: Cardiac Index
Time Frame: 24 hours post-transplant
Measure: Mean (Standard Deviation); unit: L/min/m^2
Groups:
- Standard Care Cold Storage: Patients who received standard care cold storage
- Sherpapak Cardiac Transport: Patients who received sherpapak cardiac transport
Arm/Group | Standard Care Cold Storage | Sherpapak Cardiac Transport
Number analyzed (Participants) | 10 | 10
L/min/m^2 | 3.1 (1.2) | 3.5 (1.1)

7. Secondary Outcome: Cardiac Output
Time Frame: 24 hours post-transplant
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Standard Care Cold Storage | Sherpapak Cardiac Transport
Number analyzed (Participants) | 10 | 10
L/min | 5.6 (1.3) | 6.5 (2.3)

8. Secondary Outcome: Mean Arterial Pressure
Time Frame: 24 hours post-transplant
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Standard Care Cold Storage | Sherpapak Cardiac Transport
Number analyzed (Participants) | 10 | 10
mmHg | 79 (8) | 83 (14)

9. Secondary Outcome: Pulmonary Arterial Pressure
Time Frame: 24 hours post-transplant
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Standard Care Cold Storage | Sherpapak Cardiac Transport
Number analyzed (Participants) | 10 | 10
mmHg | 25 (2) | 22 (6)

10. Secondary Outcome: Vasoactive-Inotropic Score
Description: Vasoactive inotropic scores (VIS) are used to measure the amount of cardiovascular support a patient is receiving at certain time point, for our study it was at 24hrs post transplant. Below is the calculation for the score.
  VIS = dopamine (µg/kg/min) + dobutamine (µg/kg/min) + 100 × epinephrine (µg/kg/min) + 100 × norepinephrine (µg/kg/min) + 10 × milrinone (µg/kg/min) + 10,000 × vasopressin (units/kg/min) + 50 × levosimendan (µg/kg/min).
  The minimum score is 0 if the patient does not require any support but there really isn't a maximum score as theoretically patients can be on any range of support. Higher values indicates that a patient is requiring a higher cardiovascular support at 24 hrs.
  VIS = dopamine (µg/kg/min) + dobutamine (µg/kg/min) + 100 × epinephrine (µg/kg/min) + 100 × norepinephrine (µg/kg/min) + 10 × milrinone (µg/kg/min) + 10,000 × vasopressin (units/kg/min) + 50 × levosimendan (µg/kg/min)
Time Frame: 24 hours post-transplant
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care Cold Storage | Sherpapak Cardiac Transport
Number analyzed (Participants) | 10 | 10
score on a scale | 264.1 (218) | 395.3 (418)

11. Secondary Outcome: Hospital Length of Stay
Description: Hospital Length of Stay
Time Frame: within 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard Care Cold Storage | Sherpapak Cardiac Transport
Number analyzed (Participants) | 10 | 10
days | 15.1 (8) | 21.1 (14)

12. Secondary Outcome: Acute Cellular Rejection
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care Cold Storage | Sherpapak Cardiac Transport
Number analyzed (Participants) | 10 | 10
Participants | 5 | 3

13. Secondary Outcome: 1R
Description: 1R is the rejection grade that referring to mild cellular rejection based on pathological assessment that is standardized by ISHLT. Generally, pathologist look for signs of mild cellular mediated damage (interstitial/perivascular inflammation) using special stains. Only participants with acute cellular rejection were assessed for this Outcome Measure
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care Cold Storage | Sherpapak Cardiac Transport
Number analyzed (Participants) | 5 | 3
Participants | 5 | 3

14. Secondary Outcome: Antibody Mediated Rejection
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care Cold Storage | Sherpapak Cardiac Transport
Number analyzed (Participants) | 10 | 10
Participants | 1 | 1

15. Secondary Outcome: pAMR 1
Description: pAMR1 is the rejection grade that referring to mild antibody rejection based on pathological assessment that is standardized by ISHLT. Generally, pathologist look for signs of mild antibody-mediated damage using special stains to detect the presence of immune complexes.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care Cold Storage | Sherpapak Cardiac Transport
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Within 30 days post transplant
Arm/Group | Standard Care Cold Storage | Sherpapak Cardiac Transport
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 2/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Care Cold Storage (N=10) | Sherpapak Cardiac Transport (N=10)
Epyema (Infections and infestations) | 0 | 1
Death (Cardiac disorders) | 0 | 1
Mediastinal Bleeding (Surgical and medical procedures) | 1 | 0 — Surgical complication

LIMITATIONS AND CAVEATS:
There are several limitations to our study. First, the small sample size limits our ability to detect clinical differences between the groups. Second, our primary clinical end points were only followed out to 30-days warranting further randomized trials aimed at assessing the long-term effects on clinical outcomes. Third, cardiac samples have a high dynamic range of proteins due to the abundance of contractile machinery within cardiomyocytes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT05194514/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT05194514/ICF_001.pdf